CLINICAL TRIAL: NCT01045239
Title: A Randomized, Controlled Trial Comparing Micropulse 577 nm Laser Photocoagulation And Conventional 532 nm Laser Photocoagulation for Diabetic Macular Oedema
Brief Title: Micropulse 577 nm Laser Photocoagulation Versus Conventional 532 nm Laser Photocoagulation for Diabetic Macular Oedema
Acronym: UMDMO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Assoc Prof Kenneth Choong-Sian Fong, University Malaya Eye Research Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMERC001
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Diabetic macular oedema; micropulse laser; laser treatment; macular thickness
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micropulse 577 nm yellow diode laser (Experimental)
  Interventions: Device: Micropulse 577 nm yellow diode laser
- 532 nm green diode laser (Active Comparator)
  Interventions: Device: 532 nm green diode laser

INTERVENTIONS:
Device: Micropulse 577 nm yellow diode laser — Laser administered at beginning of study and may be repeated at 16 weeks if needed
  Other Names: Quantel Supra 577nm laser
  Arms: Micropulse 577 nm yellow diode laser
Device: 532 nm green diode laser — Laser administered at beginning of study and may be repeated at 16 weeks if needed
  Arms: 532 nm green diode laser

SUMMARY:
The purpose of this study is to determine whether the new micropulse 577 nm yellow laser is a better treatment option compared to the conventional 532 nm green laser for diabetic macular edema.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a serious debilitating and deadly disease causing significant mortality and morbidity globally. Diabetic macular oedema is the most common cause of visual loss in the working population.

In 1985, the Early Treatment Diabetic Retinopathy Study (ETDRS) demonstrated that focal (direct/grid) laser photocoagulation reduces moderate vision loss from diabetic macular oedema (DMO) by 50% or more. However, further studies have shown that photocoagulation can eventually result in complications leading to loss of central vision and decreased colour vision. Thus, many newer laser machines that claim to reduce the rate of complications have been developed over the years.

In this project, we plan to evaluate the usage of the micropulse 577 nm laser, which is a yellow light laser, and compare it to the conventional 532 nm green laser that is widely used. The 577 nm laser has a high affinity for oxyhemoglobin, a slightly lower affinity for melanin and almost no affinity for macular xanthophylls, as shown in the graph below.22,23,24,25 The yellow 577 nm light also scatters very little and does not cause photochemical reactions in the tissues.

The theoretical advantage of using the micropulse 577 nm yellow laser would be the reduced energy requirement to obtain the same results as with green 532 nm. This leads to less retinal toxicity and damage due to reduced absorption by the xanthophylls. Our aim in this project is to observe whether the theoretical advantage translates to a more effective treatment in reality.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or 2)
* Diabetic macular edema in study eye associated to diabetic retinopathy
* Diffuse macular edema defined as macular thickening determined by biomicroscopy, OCT and/or fluorescein angiography.
* Best corrected visual acuity between 34 (20/200) and 68 letters (20/50).
* Macular thickness greater than 300 mcm on OCT.

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 6 months.

The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):

* Macular edema is considered to be due to a cause other than diabetic macular edema.
* Presence of vitreomacular traction.
* Concurrent proliferative diabetic retinopathy.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, significant macular ischemia, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis epiretinal membrane, or other ocular inflammatory disease, neovascular glaucoma, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of treatment for DME at any time in the past 4 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
* History of panretinal (scatter) photocoagulation (PRP) prior to enrollment or anticipated to be performed within next 6 months.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 12 months or anticipated within the next 6 months.
* History of YAG capsulotomy performed within 2 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity by logarithm of the minimum angle of resolution (LogMAR) | 1 year

SECONDARY OUTCOMES:
Macular thickness measured by optical coherence tomography (OCT) | 12 months
Photocoagulation scars on fundus photograph | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Fong, FRCOphth, Principal Investigator — University of Malaya Eye Research Centre; Tajunisah Iqbal, FRCS, Principal Investigator — University of Malaya Eye Research Centre
Locations (1):
- University Malaya Eye Research Centre, Kuala Lumpur, Malaysia